CLINICAL TRIAL: NCT00309049
Title: An Exploratory Study of Ixabepilone Administered as an Enteric Coated Formulation in Patients With Advanced Cancer.
Brief Title: Ixabepilone Administered as an Enteric Coated Formulation.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: R-Pharm (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CA163-088
Record Dates: First submitted 2006-03-29; First posted 2006-03-31 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2017-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — ixabepilone

ARMS (3):
- A1 (Active Comparator)
  Interventions: Drug: Ixabepilone
- A2 (Active Comparator)
  Interventions: Drug: Ixabepilone
- A3 (Active Comparator)
  Interventions: Drug: Ixabepilone

INTERVENTIONS:
Drug: Ixabepilone — Capsules / IV formulation, Oral/IV, 15 mg IV and 30 mg Oral (3 capsules) in cycle 1 with a sequence of IV oral and oral dosage and 40 mg IV dose every 3 weeks on cycle 2 onwards, 3 times in cycle 1 (21 days) and every 3 weeks from cycle 2 onwards, 48-96 weeks depending on response.
  Other Names: Ixempra
  Arms: A1
Drug: Ixabepilone — Capsules / IV formulation, Oral/IV, 15 mg IV and 30 mg Oral (3 capsules) in cycle 1 with a sequence of oral IV and oral dosage and 40 mg IV dose every 3 weeks on cycle 2 onwards, 3 times in cycle 1 (21 days) and every 3 weeks from cycle 2 onwards, 48-96 weeks depending on response.
  Other Names: Ixempra
  Arms: A2
Drug: Ixabepilone — Capsules / IV formulation, Oral/IV, 15 mg IV and 30 mg Oral (3 capsules) in cycle 1 with a sequence of oral oral and IV dosage and 40 mg IV dose every 3 weeks on cycle 2 onwards, 3 times in cycle 1 (21 days) and every 3 weeks from cycle 2 onwards, 48-96 weeks depending on response.
  Other Names: Ixempra
  Arms: A3

SUMMARY:
The purpose of this study is to determine the pharmacokinetics of oral Ixabepilone.

ELIGIBILITY:
Inclusion Criteria:

* ECOG status of 0-2.

Exclusion Criteria:

* Unable to swallow pills.
* Current or recent GI disease or GI surgery.
* Brain mets.
* Severe nerve damage.
* ANC <1,500/mm3
* Platelets <125K.
* Bilirubin >=1.5 times the IULN.
* ALT/AST >=1.5 times the IULN.
* Creatine >1.5 times the IULN.
* Prior treatment with Ixabepilone.
* Strong use of CYPP450 drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2006-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Determine the action of Ixabepilone in the body over a period of time including the process of absorption, distribution, metabolism and elimination.

SECONDARY OUTCOMES:
Determine the rate and extent to which Ixabepilone is absorbed or otherwise available to the treatment site in the body.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Local Institution, Washington D.C., District of Columbia
  - Local Institution, Detroit, Michigan